CLINICAL TRIAL: NCT02061592
Title: Clinical Evaluation of Two Etafilcon A Daily Disposable Lenses
Brief Title: Evaluation of Etafilcon A Daily Disposable Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5553
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etafilcon A Control Lens (Active Comparator): etafilcon A
  Interventions: Device: etafilcon A
- Etafilcon A Test Lens (Experimental): etafilcon A
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: etafilcon A
  Arms: Etafilcon A Control Lens
Device: etafilcon A
  Arms: Etafilcon A Test Lens

SUMMARY:
To evaluate the clinical performance of daily disposable etafilcon A lenses.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 and not more than 70 years of age.
* The subject's refractive cylinder must be < 1.00 Diopters (D) in each eye.
* The subject must have best corrected visual acuity of 20/25 or better in each eye.
* The subject's required spherical contact lens prescription must be in the range of -0.50 to -7.50 D in each eye.
* The subject must be a habitual and adapted wearer of daily disposable contact lenses in both eyes.
* The subject must self-report their race as Asian
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).
* The subject must demonstrate adequate mobility and 20/30 vision oculus dexter (OD) and oculus sinister (OS) with the study contact lenses.

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser in-situ keratomileusis (LASIK), etc.).
* Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Monovision or multi-focal contact lens correction.
* Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
* History of binocular vision abnormality or strabismus.
* Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self report).
* Suspicion of or recent history of alcohol or substance abuse.
* History of serious mental illness.
* History of seizures.
* Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Jacksonville, Florida
  - Honolulu, Hawaii
  - Kahului, Hawaii
  - Waipahu, Hawaii
  - ‘Aiea, Hawaii
  - New York, New York
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 128 of the 136 subjects were randomized. 8 subjects did not meet the eligibility criteria. 3 subjects were discontinued from the study. 12 subjects were excluded from analysis due to major protocol deviations. 113 subjects completed all study visits without a major protocol deviation.
Groups:
- Control/Test: Subjects first received the control lens, etafilcon A for 1 week which was to be worn for a minimum of 8 hours per day. After 1 week subjects returned for follow-up and were immediately dispensed the test lens, etafilcon A.
- Test/Control: Subjects first received the test lens, etafilcon A for 1 week which was to be worn for a minimum of 8 hours per day. Subjects then returned for follow-up and were immediately dispensed the control lens, etafilcon A
Period: Period 1
Arm/Group | Control/Test | Test/Control
Started | 66 | 62
Completed | 64 | 62
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Period 2
Arm/Group | Control/Test | Test/Control
Started | 64 | 62
Completed | 64 | 61
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consists of all randomized subjects. Randomized subjects are subjects that have signed informed consent and have been randomized to 1 of the 2 treatment arms.
Groups:
- Test/Control: Subjects first received the test lens, etafilcon A , for 1 week which was to be worn for a minimum of 8 hours per day. Subjects then returned for follow-up and were immediately dispensed the control lens, etafilcon A
- Total: Total of all reporting groups
Arm/Group | Control/Test | Test/Control | Total
Number analyzed (Participants) | 66 | 62 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (9.02) | 30.6 (7.48) | 31.0 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 66 | 62 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort
Description: Subjective assessment of comfort was performed using the Contact Lens User Experience TM (CLUE) questionnaire. CLUE was a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact lens- wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicated a more favorable/positive response with a range of 0 to 120.
Time Frame: 1-week follow-up
Population: Analysis population consisted of subjects that successfully completed the study visits without any major protocol deviations.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Subjects who received Control lens, etafilcon A, in either the first week or last week of the study.
- Test: Subjects who received the Test lens, etafilcon A, in either the first week or last week of the study.
Arm/Group | Control | Test
Number analyzed (Participants) | 113 | 113
units on a scale | 60.1 (18.47) | 43.6 (20.19)

2. Primary Outcome: Overall Vision
Description: Subjective assessment of vision was performed using the Contact Lens User Experience TM (CLUE) questionnaire. CLUE was a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact lens-wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicated a more favorable/positive response with a range of 0 to 120.
Time Frame: 1- week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test: Subjects who received Test lens, etafilcon A, in either the first week or last week of the study.
Arm/Group | Control | Test
Number analyzed (Participants) | 113 | 113
units on a scale | 64.9 (18.23) | 58.0 (19.51)

3. Primary Outcome: Monocular Logarithm of the Minimum Angle of Resolution (logMAR) Visual Acuity - Standard High Contrast Dim
Description: LogMar visual acuity within each eye was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity charts. A LogMar acuity value of 0 indicates that a subject has 20/20 vision.Positive LogMar acuity values indicate worsened vision while negative LogMar acuity values would indicated improved vision.
Time Frame: 1-week follow-up
Population: Consisted of subjects that successfully completed all study visits without any major protocol deviations. 13 Subjects were not included in the analysis population due to study procedures not properly followed from one of the investigational sites where the measured results were not collected in the lighting conditions described in the protocol.
Measure: Mean (Standard Deviation); unit: LogMar
Units Other Than Participants: Eyes
Arm/Group | Control | Test
Number analyzed (Participants) | 100 | 100
Number analyzed (Eyes) | 200 | 200
LogMar | 0.030 (0.088) | 0.020 (0.085)

4. Primary Outcome: Monocular logMar Visual Acuity - Standard Low Contrast Bright
Description: LogMar visual acuity within each eye was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity charts. A LogMar acuity value of 0 indicates that a subject has 20/20 vision. Positive LogMar acuity values indicate worsened vision while negative LogMar acuity values would indicated improved vision.
Time Frame: 1- week Follow-up
Population: Analysis population consisted of subjects that successfully completed all study visits without any major protocol deviations.
Measure: Mean (Standard Deviation); unit: LogMar
Units Other Than Participants: Eyes
Groups:
- Test: Subjects who received Test lens, etafilcon A , in either the first week or last week of the study.
Arm/Group | Control | Test
Number analyzed (Participants) | 113 | 113
Number analyzed (Eyes) | 226 | 226
LogMar | 0.060 (0.083) | 0.050 (0.079)

ADVERSE EVENTS:
Time Frame: One week for each intervention
Description: Safety Population included all subjects who were administered at least 1 test article.
Groups:
- Control: Subjects who received control lens etafilcon A in either the first or the last week of the study .
- Test: Subjects who received the test lens, etafilcon A, in either the first week or the last week of the study.
Arm/Group | Control | Test
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/113
Other Adverse Events (participants affected / at risk) | 0/113 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation the Institution will provide sponsor with at least sixty (60) days for review of a manuscript.

If needed, the Institution and Principal Investigator will withhold publication for up to an additional sixty days to allow for filing of a patent application.